CLINICAL TRIAL: NCT03848078
Title: (Cost)-Effectiveness of Optical Coherence Tomography Versus Regular Punch Biopsy in the Diagnosis and Subtyping of Basal Cell Carcinoma: a Multi Center Randomized Non-inferiority Trial
Brief Title: (Cost)-Effectiveness of Optical Coherence Tomography (OCT) in Basal Cell Carcinoma (BCC)
Acronym: ROCTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL67571.068.18; 80-85200-98-91060 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Basal Cell Carcinoma; Optical Coherence Tomography
Keywords: Basal Cell Carcinoma; Optical Coherence Tomography; Punch biopsy
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: Multi-centre randomised controlled non-inferiority trial
Who Masked: Investigator
Masking Description: The investigator is blinded for the result of the punch biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optical Coherence Tomography arm (Other): In the intervention arm, OCT imaging is performed which will take about 3 minutes. The decision on the most adequate treatment strategy will be based directly on the OCT diagnosis, but only when there is certainty about the presence of BCC and BCC subtype according to the OCT diagnosis. A 'safety' biopsy will be performed after the OCT scan. In patients where the OCT diagnosis leaves doubt or it is certain that there is no BCC, a biopsy will be taken anyway and the treatment decision will be based on the result of this punch biopsy.
  Interventions: Device: Optical Coherence Tomography
- Regular care arm (No Intervention): In patients assigned to regular care, the result of punch biopsy will always be used to decide which treatment is most adequate. Therefore, a next consultation will be planned to discuss the outcome of the biopsy and the intended treatment strategy.

INTERVENTIONS:
Device: Optical Coherence Tomography — OCT is an imaging technique, which is able to produce real-time, in vivo, cross-sectional images of lesions with a depth of 1,5-2 mm. OCT imaging is based on light-interferometry, calculating the interference of an optical beam reflected by the tissue with a reference. In such ways, microscopic details of lesions and tissues can be visualized. This information can be used to identify a lesion as BCC, and to specify the subtype. Therefore, we assume that the use of the OCT might reduce the number of biopsies and the accompanying morbidity.
  The investigator scans 6mm of skin with the OCT (30 seconds) and decides whether the lesion is a BCC or not.
  Other Names: Vivosight, Michelson diagnostics
  Arms: Optical Coherence Tomography arm

SUMMARY:
A multi-centre randomized non-inferiority trial investigating the (cost-)effectiveness of Optical Coherence Tomography (OCT) versus regular punch biopsy in the diagnosis and subtyping of Basal Cell Carcinoma (BCC).

DETAILED DESCRIPTION:
Skin cancer incidence rises worldwide due to high sun exposure and ageing. Basal cell carcinoma (BCC) is the most prevalent form, with a lifetime risk of 16-20% in the Netherlands. Currently, the gold standard for diagnosing and subtyping BCC is a punch biopsy. Since this technique is invasive, new non-invasive diagnostic methods have been developed, including optical coherence tomography (OCT). In patients with clinical and dermoscopic suspicion of BCC, OCT makes it possible to confirm and subtype BCC with high confidence, thereby obviating the need for a punch biopsy in a substantial part of patients. Hence, BCC diagnosis and treatment can be accomplished in one day. As a result, patients experience less distress and costs can be saved. By discussing diagnosis and treatment with the patient directly, care can be provided more efficiently, preventing treatment delay and saving extra hospital visits. The investigators hypothesize that the use of OCT is a cost-effective strategy when compared to regular care (always punch biopsy). However, it is important to evaluate whether an alternative OCT guided diagnostic approach does not lead to an unacceptable increase in risk of recurrent BCC.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>18 years)
* Clinical and dermoscopic suspicion of BCC
* BCC is in the differential diagnosis and a biopsy would normally be obtained to confirm the diagnosis and subtype or exclude other skin lesions.

Exclusion Criteria:

* Patients with BCC in the high-risk zone of the face (ear, nose, eye region)
* Patients with a large BCC referred to our (tertiary care) head and neck tumour working group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with treatment failure | 12 months
  The main endpoint for the non-inferiority trial is the proportion of patients with treatment failure after 12 months follow-up, where treatment failure is defined as inadequate treatment or recurrence of malignant or premalignant lesions.
Cost-effectiveness of OCT | 12 months
  The main endpoint for the cost-effectiveness analysis is the Incremental Cost-Effectiveness Ratio (ICER) defined as extra cost per gained Quality-Adjusted Life Year (QALY).

SECONDARY OUTCOMES:
The proportion of patients with avoided biopsies | 12 months
  What percentage of biopsies can be avoided in patients when using optical coherence tomography compared to regular care.
Diagnostic performance of OCT | 12 months
  The design of the study also enables evaluation of the ability of OCT to discriminate between BCC and non-BCC and between BCC subtypes (superficial, nodular and infiltrative BCC) using punch biopsy as reference standard. Diagnostic performance will be expressed as sensitivity, specificity, positive and negative predictive value. A receiver operating characteristic (ROC) curve with area under the curve (AUC) will also be calculated.
Discrete Choice Experiment to determine patient preferences | 2 months
  Patient preferences will be assessed by designing and conducting a discrete choice experiment.
Quality of life measured with EQ-5D-5L | Baseline, 12 months
  Quality of life will be evaluated using the 5-level EQ-5D version (EQ-5D-5L) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flohil SC, de Vries E, Neumann HA, Coebergh JW, Nijsten T. Incidence, prevalence and future trends of primary basal cell carcinoma in the Netherlands. Acta Derm Venereol. 2011 Jan;91(1):24-30. doi: 10.2340/00015555-1009. PMID 21264452
- [Background] Cheng HM, Guitera P. Systematic review of optical coherence tomography usage in the diagnosis and management of basal cell carcinoma. Br J Dermatol. 2015 Dec;173(6):1371-80. doi: 10.1111/bjd.14042. Epub 2015 Oct 27. PMID 26211438
- [Background] NVDV, Dutch evidence based guideline Guideline Basal Cell Carcinoma.
- [Derived] Adan F, Nelemans PJ, Essers BAB, Brinkhuizen T, Dodemont SRP, Kessels JPHM, Quaedvlieg PJF, Dermont GJ, Winnepenninckx VJL, Abdul Hamid M, Kelleners-Smeets NWJ, Mosterd K. Optical coherence tomography versus punch biopsy for diagnosis of basal cell carcinoma: a multicentre, randomised, non-inferiority trial. Lancet Oncol. 2022 Aug;23(8):1087-1096. doi: 10.1016/S1470-2045(22)00347-3. Epub 2022 Jul 11. PMID 35835136